CLINICAL TRIAL: NCT05720013
Title: Acute Effects of Beetroot Juice on Locomotor Economy and Capacity in Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, George Hornby, Professor, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 15055
Record Dates: First submitted 2022-08-22; First posted 2023-02-09 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Stroke; CVA
Keywords: dietary nitrate; Beetroot Juice; High-Intensity Gait Training
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Randomized repeated-measure crossover study
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beetroot Juice Supplement (Experimental): 140 mL of beetroot juice supplement will be ingested orally (Beet-It Nitrate 400, James White Co).
  Interventions: Dietary Supplement: Beetroot Juice supplement
- Placebo Supplement (Placebo Comparator): 140 mL of placebo supplement will be ingested orally (Beet-It Nitrate 400, James White Co).
  Interventions: Dietary Supplement: Placebo supplement

INTERVENTIONS:
Dietary Supplement: Beetroot Juice supplement — The experimental arm includes orally ingesting 140 mL Beet-It Sport Nitrate 400.
  Arms: Beetroot Juice Supplement
Dietary Supplement: Placebo supplement — he placebo arm involves orally ingesting a 140 mL placebo solution with the dietary nitrate removed.
  Other Names: Placebo Beetroot Juice supplement
  Arms: Placebo Supplement

SUMMARY:
The purpose of this study is to investigate if a beetroot juice supplement can improve oxygen capacity during walking tasks at a submaximal and maximal effort in people greater than 6 months following stroke.

DETAILED DESCRIPTION:
During this study, participants will perform baseline measurements such as walking and balance tests. During baseline testing, participants will be asked to perform a maximal exertion test while walking on a treadmill to determine the speed for a submaximal walking test. One week after baseline testing, the participant will have an intervention session where they drink either a beetroot juice supplement or a placebo. The placebo will taste similar to the beetroot juice and participants may not be able to tell the difference between the two different supplements. After a week, the participant will return to the lab and drink the other supplement. For example, if the participant drank the beetroot juice in the first session, then they will drink the placebo in the second session. During each intervention session, the participant will be asked to perform two treadmill tests, one with submaximal effort and one with maximal effort. After the walking tests, they will drink either the beetroot juice or placebo and have their blood drawn. They will wait at the hospital for 2-3 hours and have their blood drawn again. The participants will then complete the two treadmill tests again. The two intervention sessions will last about 4-6 hours for each session. Participation in the study will last 4-6 weeks including screening and baseline testing.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18-89 years
* diagnosis of chronic hemiparesis following unilateral stroke (greater than six months)
* ability to ambulate at least 0.3 m/s, with or without using an assistive device or bracing below the knee
* ability to read and understand English
* follow three-step commands

Exclusion Criteria:

* presence of cerebellar deficits
* any other neurological or orthopedic deficits that would limit walking ability
* smoking
* cannot receive physical therapy for gait-related impairments
* uncontrolled metabolic, respiratory, and cardiovascular disease

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in gait efficiency during steady state walking | Measures assessed prior to and following 2-3 hours after beetroot juice or placebo ingestion
  Oxygen Consumption during steady state walking prior to and following placebo or beetroot juice ingestion
Changes in plasma levels of Nitrate and Nitrite | Measures assessed prior to and following 2-3 hours after beetroot juice or placebo ingestion
  Blood samples taken prior and following ingestion of either the beetroot juice or placebo supplements.

SECONDARY OUTCOMES:
Changes in peak Treadmill Speed | Measures assessed prior to and following 2-3 hours after beetroot juice or placebo ingestion
  Fastest speed achieved for one minute on the treadmill during the graded treadmill test performed prior to and following placebo or beetroot juice ingestion.
Changes in peak oxygen consumption during maximum gait speed | Measures assessed prior to and following 2-3 hours after beetroot juice or placebo ingestion.
  Oxygen Consumption during maximal exertion walking during the graded treadmill test prior to and following placebo or beetroot juice ingestion
Changes in peak heart rate during the graded treadmill test | Measures assessed prior to and following 2-3 hours after beetroot juice or placebo ingestion.
  Peak heart rate during maximal exertion walking on the graded treadmill test prior to and following placebo or beetroot juice ingestion

CONTACTS AND LOCATIONS:
Locations (1):
- Rehabilitation Hospital of Indiana, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Carter SJ, Gruber AH, Raglin JS, Baranauskas MN, Coggan AR. Potential health effects of dietary nitrate supplementation in aging and chronic degenerative disease. Med Hypotheses. 2020 Aug;141:109732. doi: 10.1016/j.mehy.2020.109732. Epub 2020 Apr 9. PMID 32294579
- [Background] Coggan AR, Broadstreet SR, Mahmood K, Mikhalkova D, Madigan M, Bole I, Park S, Leibowitz JL, Kadkhodayan A, Thomas DP, Thies D, Peterson LR. Dietary Nitrate Increases VO2peak and Performance but Does Not Alter Ventilation or Efficiency in Patients With Heart Failure With Reduced Ejection Fraction. J Card Fail. 2018 Feb;24(2):65-73. doi: 10.1016/j.cardfail.2017.09.004. Epub 2017 Sep 12. PMID 28916479
- [Background] Lundberg JO, Carlstrom M, Larsen FJ, Weitzberg E. Roles of dietary inorganic nitrate in cardiovascular health and disease. Cardiovasc Res. 2011 Feb 15;89(3):525-32. doi: 10.1093/cvr/cvq325. Epub 2010 Oct 11. PMID 20937740
- [Background] Leddy AL, Connolly M, Holleran CL, Hennessy PW, Woodward J, Arena RA, Roth EJ, Hornby TG. Alterations in Aerobic Exercise Performance and Gait Economy Following High-Intensity Dynamic Stepping Training in Persons With Subacute Stroke. J Neurol Phys Ther. 2016 Oct;40(4):239-48. doi: 10.1097/NPT.0000000000000147. PMID 27632078
- [Background] Lundberg JO, Gladwin MT, Ahluwalia A, Benjamin N, Bryan NS, Butler A, Cabrales P, Fago A, Feelisch M, Ford PC, Freeman BA, Frenneaux M, Friedman J, Kelm M, Kevil CG, Kim-Shapiro DB, Kozlov AV, Lancaster JR Jr, Lefer DJ, McColl K, McCurry K, Patel RP, Petersson J, Rassaf T, Reutov VP, Richter-Addo GB, Schechter A, Shiva S, Tsuchiya K, van Faassen EE, Webb AJ, Zuckerbraun BS, Zweier JL, Weitzberg E. Nitrate and nitrite in biology, nutrition and therapeutics. Nat Chem Biol. 2009 Dec;5(12):865-9. doi: 10.1038/nchembio.260. PMID 19915529
- [Background] Lundberg JO, Weitzberg E, Gladwin MT. The nitrate-nitrite-nitric oxide pathway in physiology and therapeutics. Nat Rev Drug Discov. 2008 Feb;7(2):156-67. doi: 10.1038/nrd2466. PMID 18167491
- [Background] Coggan AR, Peterson LR. Dietary Nitrate Enhances the Contractile Properties of Human Skeletal Muscle. Exerc Sport Sci Rev. 2018 Oct;46(4):254-261. doi: 10.1249/JES.0000000000000167. PMID 30001275